CLINICAL TRIAL: NCT01282164
Title: The Diagnostic Accuracy of the Glucagon Stimulation Test for Evaluation of Adult Growth Hormone Deficiency and the Hypothalamic-Pituitary-Adrenal Axis
Brief Title: The Glucagon Stimulation Test for Evaluation of Adult Growth Hormone Deficiency and Adrenocorticotropic Axis
Acronym: GST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Massachusetts General Hospital (Other); Allegheny Endocrinology Associates (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-810
Record Dates: First submitted 2011-01-19; First posted 2011-01-24 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Adult Growth Hormone Deficiency; Hypothalamic-pituitary Disorders
Keywords: glucagon stimulation test; insulin tolerance test; growth hormone deficiency; hypothalamic-pituitary disorders
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study patients (Experimental): patients with growth hormone deficiency or hypothalamic-pituitary disorders underwent fixed-dose glucagon stimulation test (GST), weight-based GST and insulin tolerance test (ITT).
  Interventions: Procedure: Glucagon stimulation test and insulin tolerance test
- Control (Active Comparator): The control group will consist of healthy volunteers matched to the study group for age, gender, Body mass index (BMI) and estrogen status. Note: Allegheny site is not enrolling in the control group.
  Control subjects underwent fixed-dose glucagon stimulation test (GST), weight-based GST and insulin tolerance test (ITT).
  Interventions: Procedure: glucagon stimulation test and insulin tolerance test

INTERVENTIONS:
Procedure: Glucagon stimulation test and insulin tolerance test — glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test in subjects with type 2 diabetes mellitus (T2DM), coronary artery disease (CAD), cerebrovascular disease (CVD), seizure
  Arms: Study patients
Procedure: glucagon stimulation test and insulin tolerance test — glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test in subjects with type 2 diabetes mellitus (T2DM), coronary artery disease (CAD), CVD (cerebrovascular disease), seizure
  Arms: Control

SUMMARY:
The purpose of this study is to find out if the Glucagon Stimulation Test (GST) is a reliable alternative to the Insulin Tolerance Test (ITT) for diagnosis of Growth Hormone Deficiency (GHD) and adrenal insufficiency. In some patients the accuracy of the GST for evaluation of adrenal insufficiency is compared to the adrenocorticotropin hormone (ACTH ) stimulation test.

DETAILED DESCRIPTION:
Growth hormone is a protein that is produced by the pituitary gland and influences the metabolism (how fast things work) of other proteins, carbohydrates, and fats in the body. This allows the growth hormone to help humans keep a healthy balance between fat, muscle and bone throughout their life. Some people have what is called Growth Hormone Deficiency (GHD), which means that they do not produce enough growth hormone. GHD may lead to a tendency to be fat, (especially around the abdominal area), a reduced ability to exercise, heart disease, an increased possibility of breaking bones, and a general reduced quality of life.

GHD is usually evaluated through growth hormone stimulation test(s). One of the most reliable tests to evaluate if someone has GHD is by using arginine + Growth Hormone Releasing Hormone (GHRH) test. However, Since 2008 GHRH is no longer available in the USA. For this reason there has been a significant gap for an alternative test for evaluation of patients suspected to have GHD that can be easily performed and be reliable. The Insulin Tolerance Test (ITT) is generally considered the gold standard test for evaluation of growth hormone (GH) deficiency. The ITT involves giving insulin intravenously (through a plastic tube inserted in your vein) to lower your blood sugar followed by the collection of blood samples to evaluate how your body handles low blood sugar. There are side effects of the ITT including hypoglycemia (low blood sugar causing you to become weak, perspire, shaky and have some mental cloudiness) which can be unpleasant. ITT can not be performed in patients older than 65 years of age and in those with certain medical conditions such as history of heart disease, seizure disorder or stroke. At the same time, the ITT needs to be done by an experienced clinician and requires trained staff to perform. For this reason there is a need for an alternative reliable test for evaluation of GHD.

The second purpose of this study is to find out if you have adrenal insufficiency. Cortisol is a hormone produced by the adrenal gland and is released in response to stress. Cortisol production is regulated through the hypothalamus and the pituitary gland. Its primary functions are to increase blood sugar, regulate the immune system and aid in fat, protein and carbohydrate metabolism. Patients with low cortisol may experience fatigue, body ache, sleep disturbance, nausea and mood changes. Pituitary disorders may lead to low cortisol levels and can cause symptoms associated with adrenal insufficiency. The Insulin Tolerance Test (ITT) can also be used for the evaluation of adrenal function. Patients who can not undergo ITT, can be evaluated by the ACTH (adrenocorticotropic hormone) Stimulation Test, which is generally very well tolerated. Preliminary results from previous studies indicate that the Glucagon Stimulation Test (GST) may be used to evaluate adrenal function. The investigators in this study will compare your cortisol levels during two different GSTs with the cortisol levels achieved during ITT or ACTH stimulation test.

Since the 1970s, the Glucagon Stimulation Test (GST) has been used by several research studies for evaluation of GHD and adrenal insufficiency. Glucagon is a hormone produced in the pancreas and is secreted during times of low blood sugar or in response to growth hormone. It is used to raise very low blood sugar and in diagnostic testing of the stomach and other digestive organs. Glucagon is readily available, relatively inexpensive and generally well tolerated; the major side effects include upset stomach that can lead to vomiting and headaches. It can be used in patients with diabetes and those older than 65 years of age.

The glucagon stimulation test (GST) has been suggested as an alternative test to ITT for evaluation of growth hormone deficiency (GHD) and adrenal insufficiency. The test is similar to the ITT and ACTH Stimulation Test in that blood samples are taken both before and after the medication is given. Glucagon is given intramuscularly (as in injection in your muscle). The fewer side effects make this an attractive substitute for the ITT. The 2007 consensus guideline by the GH Research Society considers GST as a test that may be used for evaluation of patients suspected to have GHD. However, the same statement does not provide any diagnostic cut-off value for GH during the GST. The purpose of this study is to see if the GST can be an accurate substitute for the ITT in the evaluation of both GHD and adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* male and female
* hypothalamic pituitary disorders (study subjects)
* history of regular, age appropriate menses (control subjects)
* male subjects with normal serum testosterone and follicle stimulating hormone (FSH) (control subjects)
* normal FSH in post-menopausal subjects (control subjects)
* normal thyroid stimulating hormone (TSH), free thyroxine (T4), prolactin (control subjects)

Exclusion Criteria:

* unable to give consent
* pregnancy
* active acromegaly
* pheochromocytoma
* active Cushing's disease
* pituitary insult within past 6 weeks
* elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
* renal failure
* history of malignancy
* severe acute illness
* uncontrolled hypertension
* Diabetes mellitus (DM) type 1
* Hemoglobin (Hgb) A1c >9% in last 3 months in Type 2 DM
* severe coronary artery disease
* women <50 years of age with untreated hypogonadism
* men with untreated hypogonadism
* growth hormone treatment in the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hamrahian, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic Endocrinology, Diabetes and Metabolism, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 patients with hypothalamic-pituitary disorders and 1-2 (n = 14) or 3 or more (n = 14) pituitary hormone efficiencies (PHD) were recruited from four pituitary centers.
  A control group of 14 subjects was also recruited and underwent the insulin tolerance test (ITT) and the two glucagon stimulation tests (GSTs).
Pre-assignment Details: There was no wash out period. Patients and controls were eligible for the study after the initial office visit for eligibility criteria, signing the consent form followed by labs to make sure that they are eligible for the study. One patient was excluded since the patient did not achieve hypoglycemia during insulin tolerance test
Groups:
- Study Patients: patients with growth hormone deficiency or hypothalamic-pituitary disorders
  Glucagon stimulation test and insulin tolerance test: glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg adrenocorticotropin hormone (ACTH) stimulation test in subjects with type 2 diabetes mellitus (T2DM), coronary artery disease (CAD), cerebrovascular disease (CVD), seizure
- Control: The control group will consist of healthy volunteers matched to the study group for age, gender, BMI and estrogen status. Note: Allegheny site is not enrolling in the control group.
  glucagon stimulation test and insulin tolerance test: glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test in subjects with T2DM, CAD, CVD, seizure
Period: Overall Study
Arm/Group | Study Patients | Control
Started | 29 | 14
Completed | 28 | 14
Not Completed | 1 | 0
Not completed — Lack of hypoglycemia during ITT | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient did not achieve hypoglycemia during the insulin tolerance test
Groups:
- Study Patients: patients with growth hormone deficiency or hypothalamic-pituitary disorders
  Glucagon stimulation test and insulin tolerance test: glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test in subjects with T2DM, CAD, CVD, seizure
- Total: Total of all reporting groups
Arm/Group | Study Patients | Control | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 14 | 39
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (11.9) | 49.0 (12.2) | 50.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 14 | 6 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Peak GH Level in Adult Patients With Hypothalamic-pituitary Disorders and 1-2 Pituitary Hormone Deficiency (PHD).
Description: The peak growth hormone (GH) during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in patients with adult onset hypothalamic-pituitary disease and 1-2 pituitary hormone deficiency (PHD) other than growth hormone (GH) deficiency.
Time Frame: one year
Population: Peak GH levels during Insulin Tolerance test, fixed-dose GST and weight-based GST in Patients with hypothalamic-pituitary disorders and 1-2 pituitary hormone deficiency other than GH deficiency. One patient older than 65 years underwent adrenocorticotropin hormone (ACTH) stimulation test instead of ITT.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Patients With 1-2 PHD- Insulin Tolerance Test: Patients with hypothalamic-pituitary disorders and 1-2 pituitary hormone deficiency (PHD) other than GH deficiency
  insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test was used in 3 subjects who were not eligible for ITT
- Patients With 1-2 PHD- Fixed Dose GST; Patients With 1-2 PHD- Weight Based GST: Patients with hypothalamic-pituitary disorders and 1-2 pituitary hormone deficiency (PHD) other than GH deficiency
Arm/Group | Patients With 1-2 PHD- Insulin Tolerance Test | Patients With 1-2 PHD- Fixed Dose GST | Patients With 1-2 PHD- Weight Based GST
Number analyzed (Participants) | 13 | 14 | 14
ng/mL | 0.9 [0.2 to 18.8] | 0.6 [0.1 to 6.9] | 0.7 [0.1 to 11.7]

2. Primary Outcome: Peak Growth Hormone (GH) Level in Healthy Volunteers
Description: The peak growth hormone (GH) during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in healthy volunteers
Time Frame: one year
Measure: Median (Full Range); unit: ng/mL
Groups:
- Control Group- ITT: The control group consist of healthy volunteers matched to the study group for age, gender, BMI and estrogen status. Note: Allegheny site did not enroll the control group. All underwent insulin tolerance test using 0.10-0.15 U/kg
- Control Group- Fixed-dose GST; Control Group- Weight-based GST: The control group consist of healthy volunteers matched to the study group for age, gender, BMI and estrogen status. Note: Allegheny site is not enrolling in the control group.
Arm/Group | Control Group- ITT | Control Group- Fixed-dose GST | Control Group- Weight-based GST
Number analyzed (Participants) | 14 | 14 | 14
ng/mL | 14.0 [2.5 to 42.7] | 4.5 [1.3 to 11.3] | 5.8 [2.3 to 24.5]

3. Primary Outcome: Peak GH Level in Adult Patients With Hypothalamic-pituitary Disorders and Three or More Pituitary Hormone Deficiency (PHD).
Description: The peak growth hormone (GH) during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in patients with adult onset hypothalamic-pituitary disease with three or more pituitary hormone deficiency (PHD) other than growth hormone (GH) deficiency.
Time Frame: one year
Population: Peak GH levels during Insulin Tolerance test, fixed-dose GST and weight-based GST in Patients with hypothalamic-pituitary disorders with three or more pituitary hormone deficiency other than GH deficiency. Two patients older than 65 years underwent adrenocorticotropin hormone (ACTH) stimulation test instead of ITT.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Patients With 3 or More PHD- Insulin Tolerance Test: Patients with hypothalamic-pituitary disorders and three or more pituitary hormone deficiency (PHD) other than GH deficiency
  insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test was used in 3 subjects who were not eligible for ITT
- Patients With 3 or More PHD- Fixed Dose GST; Patients With 3 or More PHD- Weight Based GST: Patients with hypothalamic-pituitary disorders and three or more pituitary hormone deficiency (PHD) other than GH deficiency
Arm/Group | Patients With 3 or More PHD- Insulin Tolerance Test | Patients With 3 or More PHD- Fixed Dose GST | Patients With 3 or More PHD- Weight Based GST
Number analyzed (Participants) | 12 | 14 | 14
ng/mL | 0.1 [0.1 to 4.4] | 0.1 [0.1 to 2.8] | 0.1 [0.1 to 2.1]

4. Primary Outcome: Peak Cortisol Level in Adult Patients With Hypothalamic-pituitary Disorders and 1-2 Pituitary Hormone Deficiency (PHD).
Description: The peak cortisol level during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in patients with adult onset hypothalamic-pituitary disease and 1-2 pituitary hormone deficiency (PHD) other than growth hormone (GH) deficiency.
Time Frame: one year
Population: Peak cortisol levels during Insulin Tolerance test, fixed-dose GST and weight-based GST in Patients with hypothalamic-pituitary disorders and 1-2 pituitary hormone deficiency other than GH deficiency. One patient older than 65 years of age underwent ACTH stimulation test instead of ITT
Measure: Median (Full Range); unit: ug/dL
Arm/Group | Patients With 1-2 PHD- Insulin Tolerance Test | Patients With 1-2 PHD- Fixed Dose GST | Patients With 1-2 PHD- Weight Based GST
Number analyzed (Participants) | 13 | 14 | 14
ug/dL | 22.2 [18.6 to 29.3] | 19.5 [12.5 to 32.4] | 22.7 [15.4 to 32.2]

5. Primary Outcome: Peak Cortisol Level in Healthy Volunteers.
Description: The peak cortisol levels during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in healthy volunteers.
Time Frame: one year
Population: Peak cortisol levels during Insulin Tolerance test, fixed-dose GST and weight-based GST in healthy volunteers
Measure: Median (Full Range); unit: ug/dL
Arm/Group | Control Group- ITT | Control Group- Fixed-dose GST | Control Group- Weight-based GST
Number analyzed (Participants) | 14 | 14 | 14
ug/dL | 22.1 [18.1 to 28.5] | 18.0 [11.5 to 26.7] | 22.7 [13.8 to 31.4]

6. Primary Outcome: Peak Cortisol Level in Adult Patients With Hypothalamic-pituitary Disorders and Three or More Pituitary Hormone Deficiency (PHD).
Description: The peak cortisol level during Insulin Tolerance Test (ITT), fixed- dose glucagon stimulation test (GST) and weight-based GST in patients with adult onset hypothalamic-pituitary disease and three or more pituitary hormone deficiency (PHD) other than growth hormone (GH) deficiency.
Time Frame: one year
Population: Peak cortisol level during Insulin Tolerance test, fixed-dose GST and weight-based GST in Patients with hypothalamic-pituitary disorders with three or more pituitary hormone deficiency other than GH deficiency. Two patients older than 65 years of age underwent adrenocorticotropin hormone (ACTH) stimulation test instead of ITT.
Measure: Median (Full Range); unit: ug/dL
Arm/Group | Patients With 3 or More PHD- Insulin Tolerance Test | Patients With 3 or More PHD- Fixed Dose GST | Patients With 3 or More PHD- Weight Based GST
Number analyzed (Participants) | 12 | 14 | 14
ug/dL | 6.3 [1.0 to 18.0] | 2.3 [1.0 to 16.9] | 2.5 [1.0 to 19.7]

7. Primary Outcome: Peak Cortisol Level During Adrenocorticotropin Hormone (ACTH) Stimulation Test
Description: The peak cortisol level during ACTH stimulation test in 3 patients with adult onset hypothalamic-pituitary disease who were older than 65 years of age and could not under go insulin tolerance test (ITT).
Time Frame: one year
Population: Peak cortisol level during ACTH stimulation test in three patients with hypothalamic-pituitary disorders who were older than 65 and could not undergo ITT based on the study protocol
Measure: Median (Full Range); unit: ug/dL
Groups:
- Patients Older Than 65: Three patients with adult onset hypothalamic-pituitary disease underwent who were older than 65 years of age underwent ACTH stimulation test instead of ITT.
Arm/Group | Patients Older Than 65
Number analyzed (Participants) | 3
ug/dL | 10 [1.2 to 23.5]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Observation during dynamic testing and follow up telephone call
Groups:
- Study Patients: patients with hypothalamic-pituitary disorders
  Glucagon stimulation test and insulin tolerance test: glucagon stimulation test using 1 mg (1.5 mg if weigh >90 kg) glucagon stimulation test using 0.03 mg/kg (maximum dose 3 mg) insulin tolerance test using 0.10-0.15 U/kg ACTH stimulation test in subjects with T2DM, CAD, CVD, seizure
Arm/Group | Study Patients | Control
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/14
Other Adverse Events (participants affected / at risk) | 16/28 | 9/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Patients (N=28) | Control (N=14)
Nausea (Gastrointestinal disorders) | 10 (13) | 5 (9)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (2)
Headache (Nervous system disorders) | 2 (3) | 1 (2)
Dizziness (Nervous system disorders) | 2 (3) | 2 (3)

LIMITATIONS AND CAVEATS:
This includes the relatively small number of subjects, and that the majority of patients had growth hormone deficiency (GHD), so a larger study assessing adults with mild hypothalamic-pituitary disease and possible but unconfirmed GHD is required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No